CLINICAL TRIAL: NCT00309660
Title: Treatment With Local PPARgamma Ligand in Distal Ulcerative Colitis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Herlev Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PPAR2005
Record Dates: First submitted 2006-03-30; First posted 2006-04-03 (Estimated); Last update posted 2006-09-21 (Estimated); Status verified 2006-09

CONDITIONS: Ulcerative Colitis
Keywords: PPARgamma ligand; Rosiglitazone; Enema
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Rosiglitazone

INTERVENTIONS:
Drug: Rosiglitazone

SUMMARY:
Treatment with PPARgamma ligands have been shown to reduces intestinal inflammation in murine models of colitis. The aim of this study was to evaluate the effect of treatment with local PPARgamma ligand (rosiglitazone) in distal ulcerative colitis.The patients are treated with rosiglitazone enema, once a day, for fourteen days. Disease activity was assessed before and after treatment by endoscopical and clinical activity score.

ELIGIBILITY:
Inclusion Criteria:

* Distal ulcerative colitis (Mayo Clinical Score > 7)
* Age > 18 years
* Written consent

Exclusion Criteria:

* Age < 18 years
* Severe ulcerative colitis
* Systemic treatment with steroids or azathioprin within the last 3 month
* Known liver or kidney disease
* Severe heart failure
* Pregnancy or breast feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-11; Study Completion 2007-06

PRIMARY OUTCOMES:
Clinical response

SECONDARY OUTCOMES:
Endoscopic response

CONTACTS AND LOCATIONS:
Overall Officials: Jørn Brynskov, Ass. Prof., Principal Investigator — Dept Gastroenterology C, Herlev University Hospital, 2730 Herlev, Denmark
Locations (1):
- Dept. Gastroenterology C, Herlev University Hospital, Herlev, Denmark